CLINICAL TRIAL: NCT03878849
Title: Phase 2, Randomized, Prospective, Open-Label, Parallel-Arm, Dose Optimization Study to Investigate the Safety, Tolerability, PK/PD, and Anti- Tumor Effect of 2X-121 in Patients With Recurrent, Advanced Ovarian Cancer.
Brief Title: Investigation of the Anti-tumor Effect of 2X-121 in Patients With Recurrent, Advanced Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Allarity Therapeutics (Industry)
Collaborators: Alcedis GmbH (Industry); Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (PARPi) 2X-1002; 2020-000539-31 (EudraCT Number)
Record Dates: First submitted 2019-03-08; First posted 2019-03-18 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Advanced Ovarian Cancer
MeSH Terms: interventions — stenoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: 2X-121 600 mg (Experimental): 2X-121 will be administered daily as 600 mg (200 mg 2X-121 morning dose + 400 mg (2 x 200 mg) 2X-121 evening dose) hard gelatin capsules in a 28 days cycle.
  Interventions: Drug: 2X-121
- Drug: 2X-121 800 mg (Experimental): 2X-121 will be administered 800 mg (400 mg (2 x 200 mg) 2X-121 morning dose + 400 mg (2 x 200 mg) 2X-121 evening dose) hard gelatin capsules in a 28 days cycle.
  Interventions: Drug: 2X-121

INTERVENTIONS:
Drug: 2X-121 — 2X-121 will be administered daily as 600 mg (200 mg 2X-121 morning dose + 400 mg (2 x 200 mg) 2X-121 evening dose) hard gelatin capsules in a 28 days cycle.
  Other Names: E7449, MGI25036
  Arms: Drug: 2X-121 600 mg
Drug: 2X-121 — 2X-121 will be administered daily as 800 mg (400 mg (2 x 200 mg) 2X-121 morning dose + 400 mg (2 x 200 mg) 2X-121 evening dose) hard gelatin capsules in a 28 days cycle.
  Arms: Drug: 2X-121 800 mg

SUMMARY:
The purpose of this study is to evaluate the optimal dose of 2X-121 as single agent therapy at 600 mg daily (split BID 200 mg morning + 400 mg evening) compared to 800 mg daily (split BID 400 mg morning + 400 mg evening) in recurrent, advanced ovarian cancer patients that have platinum-resistant disease, defined as progression within 6 months after the last dose of platinum-based chemotherapy, or are platinum ineligible. The optimal dose will be selected based on an integrated analysis of PK/PD, safety, and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Age 18 years or older.
3. Histologically or cytologically documented epithelial ovarian, fallopian tube, or primary peritoneal tumors, with high-grade serous or endometrioid, or predominantly serous/endometrioid histology (independent of BRCA1 and HRD status).
4. Patients must have platinum-resistant disease, defined as progression within 6 months after the last dose of platinum-based chemotherapy, or are platinum ineligible.
5. Patients have received no more than one line of therapy in the platinum resistant or platinum ineligible setting. Note: Prior ADCs therapy (e.g., Elahere) will not count towards this previous line of therapy.
6. Measurable disease by CT scan or MRI. Note: Baseline tumor assessment will be performed within 4 weeks prior to Day 1 Cycle 1
7. Performance status of ECOG ≤ 1.
8. Patients must have a life expectancy of >16 weeks.
9. Recovered to Grade 1 or less from prior surgery or acute toxicities of prior radiotherapy, or treatment with cytotoxic, hormonal, or biologic agents.
10. Adequate conditions as evidenced by the following clinical laboratory values:

    1. Absolute neutrophils count (ANC) ≥ 1.5 x 103 μL
    2. Hemoglobin > 9.0 g/dL
    3. Platelets ≥ 100 x 103 μL
    4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase ≤ 2.5 x ULN, unless liver metastases are present, in which case they must be ≤5 x ULN
    5. Serum bilirubin ≤ 1.5 ULN
    6. Creatinine ≤ 1.5 ULN
    7. Blood urea nitrogen (BUN) ≤2X ULN.
11. FFPE tumor tissue should be available from the current relapse, if obtainable, otherwise the most recent archival tumor tissue. Note: Patients treated with a PARP inhibitor must have a new biopsy unless there is an archival biopsy that was done after the PARP inhibitor treatment was discontinued.
12. Negative serum pregnancy test in women of childbearing potential (WOCBP). WOCBP is defined as premenopausal women or less than 12 months of amenorrhea post-menopause, and women who have not undergone surgical sterilization or hysterectomy or bilateral salpingo-oophorectomy.
13. Sexually active females of childbearing potential must use adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception) for the study duration and at least six months afterwards.

Exclusion Criteria:

1. Patients who have platinum-refractory disease, defined as progression during the last platinum-based chemotherapy.
2. Concurrent chemotherapy, antibody therapies radiotherapy,hormonal therapy, or other investigational drug except non-disease related conditions (e.g. insulin for diabetes) during study period.
3. Other malignancy with exception of any stage I and II cancer that is deemed cured by the Investigator.
4. Any active infection requiring parenteral or oral antibiotic treatment.
5. Known HIV positivity.
6. Known active hepatitis B or C.
7. Clinically significant cardiovascular disease:

   1. Stroke within ≤ 12 months prior to day 1
   2. Transient ischemic attach (TIA) within ≤ 12 months prior to day 1
   3. Myocardial infarction within ≤ 12 months prior to day 1
   4. Unstable angina
   5. New York Heart Association (NYHA) Class II or greater congestive heart failure (CHF)
   6. Uncontrolled cardiac arrhythmia requiring medication
8. Other medications or conditions that in the Investigator's opinion would contraindicate study participation for safety reasons or interfere with the interpretation of study results.
9. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of 2X-121.
10. Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy.
11. Patients unable to be regularly followed for any reason (geographic, familiar, social, psychological, housed in an institution e.g., prison because of a court agreement or administrative order).
12. Patients, who are close colleagues, associates, or family members of, or in any way dependent on the sponsor or the investigator.
13. Ascites requiring drainage >500cc in the 2 weeks prior to enrolment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the optimal dose of 2X-121 as single agent therapy | From enrollment up to approximately 2 years
  To evaluate the optimal dose of 2X-121 as single agent therapy at 600 mg daily compared to 800 mg daily.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | From enrollment up to approximately 2 years
Progression free survival | From enrollment up to approximately 2 years
Overall survival | From enrollment up to approximately 2 years
Evaluate disease control rate (DCR) | At baseline and start of each cycle, up to approximately 2 years
Evaluate objective response rate (ORR) | From enrollment up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - OU Health Stephenson Cancer, Oklahoma City, Oklahoma
  - Swedish Center for Research and Innovation, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No